CLINICAL TRIAL: NCT03300752
Title: Self-care Decision-making: Feasibility of the BREATHE Asthma Intervention Trial - Phase II (Part 2 - a Pilot Randomized Trial Phase)
Brief Title: Validation of the BREATHE Asthma Intervention Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Maureen George, Associate Professor of Nursing at the Columbia University Medical Center, Nursing Scholarship & Research, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: AAAR5216
Record Dates: First submitted 2017-09-29; First posted 2017-10-03 (Actual); Results first posted 2021-09-28 (Actual); Last update posted 2021-09-28 (Actual); Status verified 2021-09

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BREATHE Intervention (Experimental): The patient's primary care provider (PCP) will deliver the active intervention (shared decision-making discussion of asthma control status and treatment) - BREATHE Intervention.
  Interventions: Behavioral: BREATHE Intervention
- Control Intervention (Active Comparator): The patient's primary care provider (PCP) will deliver the control intervention (discussion of healthy lifestyles).
  Interventions: Behavioral: Control Intervention

INTERVENTIONS:
Behavioral: BREATHE Intervention — PCPs randomized to BREATHE will receive the tablet which, when the screen is advanced by the PCP, will prompt the PCP through a 7-minute, 4-step brief intervention tailored to respond to the patient's specific beliefs, and shared decision-making discussion of asthma control status and treatment.
  Arms: BREATHE Intervention
Behavioral: Control Intervention — PCP will provide discussion of healthy lifestyles.
  Arms: Control Intervention

SUMMARY:
The overall goal of this study to preliminarily validate a novel intervention delivered by primary care providers (PCPs) to their Black adult patients with uncontrolled asthma in federally qualified health centers (FQHCs).

DETAILED DESCRIPTION:
Nearly every asthma related hospitalization and death could be prevented with appropriate self-management that achieves and maintains disease control. However, as many as 64% of adults have uncontrolled asthma; minorities are disproportionately represented within that population. While inhaled corticosteroids (ICS) are a safe and effective treatment for uncontrolled asthma, relative to Whites, Blacks have lower rates of ICS adherence.

Black adults with uncontrolled asthma experience profound health disparities. Despite data that point to the critical need for enhanced asthma self-management, rates of controlled asthma are well below Healthy People 2020 targets, particularly among vulnerable populations. This Brief Evaluation of Asthma Therapy (BREATHE) intervention has the potential to offer a new avenue to asthma control via shared decision-making that supports ICS adherence.

ELIGIBILITY:
PROVIDER RECRUITMENT

Inclusion Criteria:

* PCPs (MDs and Nurse Practitioners (NPs)/Physician Assistants (PAs)) working in family, primary or internal medicine care services
* Who have at least 40 adult patients with persistent asthma (defined as having been prescribed ICS) on their patient panel

Exclusion Criteria:

* PCPs whose primary focus is outside of adult health services (family, primary or internal medicine), such as behavioral health, pediatrics and Obstetrics and Gynaecology (OB-GYN)

PATIENT RECRUITMENT

Inclusion Criteria:

Patients must be

1. adults (> or = 18 years of age) who self-report race as Black or African American
2. with PCP-diagnosed persistent asthma
3. prescribed ICS
4. receiving asthma care at participating FQHCs
5. who have uncontrolled asthma
6. have erroneous personal health and/or negative ICS beliefs

Exclusion Criteria:

1. participation in Phase 1 (Part 1) of the BREATHE trial (focus groups)
2. non-English speaking
3. serious mental health conditions (e.g., psychosis) that preclude completion of study procedures or confound analyses

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2019-05-29 (Actual); Study Completion 2019-05-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maureen George, PhD, Principal Investigator — Associate Professor of Nursing at Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] George M, Pantalon MV, Sommers MLS, Glanz K, Jia H, Chung A, Norful AA, Poghosyan L, Coleman D, Bruzzese JM. Shared decision-making in the BREATHE asthma intervention trial: A research protocol. J Adv Nurs. 2019 Apr;75(4):876-887. doi: 10.1111/jan.13916. Epub 2019 Jan 24. PMID 30479020
- [Derived] George M, Bruzzese JM, Lynn S Sommers M, Pantalon MV, Jia H, Rhodes J, Norful AA, Chung A, Chittams J, Coleman D, Glanz K. Group-randomized trial of tailored brief shared decision-making to improve asthma control in urban black adults. J Adv Nurs. 2021 Mar;77(3):1501-1517. doi: 10.1111/jan.14646. Epub 2020 Nov 29. PMID 33249632

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | BREATHE Intervention | Control Intervention
Started | 40 | 40
Completed | 38 | 38
Not Completed | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | BREATHE Intervention | Control Intervention | Total
Number analyzed (Participants) | 40 | 40 | 80
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.35 (12.80) | 42.9 (13.06) | 45.1 (13.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 36 | 66
  Male | 10 | 4 | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 38 | 35 | 73
  White | 0 | 0 | 0
  More than one race | 2 | 5 | 7
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 40 | 40 | 80

OUTCOME MEASURES:

1. Primary Outcome: Asthma Control Questionnaire (ACQ) Score
Description: Full title: Asthma Control Questionnaire Construct measured: self-reported asthma control Scoring: 0 points = total asthma control/ best outcome, 6 points = completely uncontrolled asthma/ worst outcome
Time Frame: Baseline, 1 Month, 2 Months, 3 Months (post-intervention)
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | BREATHE Intervention | Control Intervention
Number analyzed (Participants) | 40 | 40
score on a scale
  Baseline | 2.94 (0.15) | 2.63 (0.15)
  1-month post | 2.17 (0.17) | 2.16 (0.16)
  2-month post | 2.22 (0.16) | 2.35 (0.16)
  3-month post | 2.40 (0.15) | 2.24 (0.15)

2. Secondary Outcome: Asthma Quality of Life Questionnaire (AQLQ) Score
Description: Full title: Asthma Quality of Life Questionnaire Construct: quality of life for patients with asthma Scoring: 32 items, each scored 1-7. The total score is calculated as a mean of all 32 items (1= low quality of life/ worse outcome, 7= high quality of life/ best outcome)
Time Frame: Baseline, 1 Month, 2 Months, 3 Months (post-intervention)
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | BREATHE Intervention | Control Intervention
Number analyzed (Participants) | 40 | 40
score on a scale
  Baseline | 3.50 (0.18) | 3.65 (0.18)
  1-month post | 4.03 (0.20) | 4.07 (0.19)
  2-month post | 3.97 (0.19) | 4.18 (0.19)
  3-month post | 4.02 (0.18) | 4.22 (0.18)

3. Secondary Outcome: Medication Adherence Record Scale-Asthma (MARS-A) Score
Description: Full title: Medication Adherence Record Scale- Asthma Construct: Adherence to inhaled corticosteroid medications Scoring: Total score is calculated as a mean of the 10 items, scores range from 1-5 (1= low adherence/ worse outcome, 5= high adherence/ best outcome)
Time Frame: Baseline, 1 Month, 2 Months, 3 Months (post-intervention)
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | BREATHE Intervention | Control Intervention
Number analyzed (Participants) | 40 | 40
score on a scale
  Baseline | 3.95 (0.12) | 3.88 (0.12)
  1-month post | 4.07 (0.13) | 4.12 (0.12)
  2- month post | 4.28 (0.12) | 4.18 (0.12)
  3-month post | 4.08 (0.12) | 4.03 (0.12)

ADVERSE EVENTS:
Time Frame: Up to 3 months post-intervention
Arm/Group | BREATHE Intervention | Control Intervention
All-Cause Mortality (participants affected / at risk) | 1/40 | 1/40
Serious Adverse Events (participants affected / at risk) | 1/40 | 0/40
Other Adverse Events (participants affected / at risk) | 5/40 | 2/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BREATHE Intervention (N=40) | Control Intervention (N=40)
presumed myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) — The participant experienced a sudden unexplained death at home. The family reported that the participant's clinician attributed it as likely "a heart attack'
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BREATHE Intervention (N=40) | Control Intervention (N=40)
emergency department visit (Respiratory, thoracic and mediastinal disorders) | 5 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-08): https://cdn.clinicaltrials.gov/large-docs/52/NCT03300752/Prot_SAP_000.pdf